CLINICAL TRIAL: NCT00607321
Title: The Medtronic Bare Metal Bifurcation Stent Clinical Trial in Humans
Brief Title: Bare Metal Bifurcation Stent Clinical Trial in Humans
Acronym: BRANCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP088
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Results first posted 2011-08-31 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
Keywords: restenosis; Coronary Disease; Coronary Arteriosclerosis; Arterial Occlusive Diseases
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Medtronic Bifurcation Stent System
  Interventions: Device: Medtronic Bifurcation Stent System

INTERVENTIONS:
Device: Medtronic Bifurcation Stent System — Percutaneous Coronary Stenting

SUMMARY:
To assess the feasibility and safety of the Medtronic Bifurcation Stent System for the treatment of single de novo bifurcation lesions in native coronary arteries with reference vessel diameters (RVD) for the proximal main vessel of 3.8 - 4.3 mm, distal main branch of 3.0 - 3.5 mm, and side branch RVD up to 2.5 mm.

ELIGIBILITY:
General Inclusion Criteria

* Candidate for percutaneous coronary intervention & emergent coronary artery bypass graft surgery
* Clinical evidence of ischemic heart disease or a positive functional study
* Female patients of childbearing potential has negative pregnancy test within 7 days before trial procedure
* Patient or patient's legal representative provided written informed consent
* Patient agrees to comply with follow-up evaluations

Angiographic Inclusion Criteria

* Target lesion ia a single de novo bifurcation lesion involving a native coronary artery with reference vessel diameter for the proximal main of 3.8 - 4.3 mm, distal main of 3.0 - 3.5 mm, & side branch RVD up to 2.5 mm
* Acceptable target lesion lengths are any combination of:
* <16mm proximally from carina in proximal main vessel
* <16mm distally from the carina in distal main branch
* <12mm from carina in side branch
* Target lesion in main vessel has stenosis of > 50% and <100%
* Target vessel has (TIMI) flow >2

General Exclusion Criteria

* Known hypersensitivity/contraindication to aspirin, heparin or bivalirudin, clopidogrel or ticlopidine, cobalt, nickel, chromium, molybdenum, or sensitivity to contrast media, which can't be adequately pre-medicated
* Platelet count <100,000 cells/mm³ or >700,000 cells/mm³, or a white blood cell (WBC) count <3,000 cells/mm³ within 7 days prior to index procedure
* Serum creatinine level >170 micromol/L within 7 days prior to index procedure
* Evidence of acute MI within 72 hours of intended trial procedure (defined as: QWMI or NQWMI having CK enzymes >2X laboratory upper limit of normal with presence of elevated CK-MB (any amount above laboratory upper limit of normal)
* Previous stenting anywhere in target vessel
* PCI of non-target vessel within 30 days prior to procedure that results in any MACE event. If non target vessel stent is implanted within 72 hours prior to index procedure, 2 post procedural serial CK or CK-MB measurements must be below investigational site's upper limit of normal.
* PCI of non-target vessel within 24 hours prior to procedure
* Planned PCI of any vessel within 30 days post-procedure
* Planned PCI of the target vessel within 6 months post-procedure
* During index procedure, target lesion requires treatment with device other than PTCA or cutting balloon prior to stent placement
* Documented left ventricular ejection fraction (LVEF) <30% at most recent evaluation.
* History of stroke or transient ischemic attack (TIA) within prior 6 months
* Active peptic ulcer or upper gastrointestinal (GI) bleeding within prior 6 months
* History of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Concurrent medical condition with life expectancy < 12 months
* Currently participating in investigational drug or device trial that's not completed the primary endpoint or that clinically interferes with current trial endpoints; or requires coronary angiography, IVUS or other coronary artery imaging procedures.

Angiographic Exclusion Criteria

* Bifurcation angle of >90 degrees by visual estimate
* Target lesion located in native vessel with saphenous vein graft or left/right internal mammary artery (LIMA/RIMA) bypass
* Significant stenosis (>50%) proximal or distal to target lesion that might require revascularization or impede run off.
* Target vessel is excessively tortuous (two bends >90º to reach target lesion)
* Target lesion has any of following characteristics:
* Lesion location is aorto-ostial, unprotected left main lesion, or within 5 mm of origin of left anterior descending (LAD), left circumflex (LCX), or right coronary artery (RCA).
* Severely calcified
* Evidence of thrombus
* Co-existence of unprotected left main coronary artery disease (obstruction >50% in left main coronary artery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Meredith, MD, Principal Investigator — Monash Medical Centre
Locations (1):
- Auckland City Hospital, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Groups:
- Medtronic Bifurcation Stent System: Single arm, All patients single de novo bifurcation lesions; 7 run-in subjects not included in analysis
Period: Overall Study
Arm/Group | Medtronic Bifurcation Stent System
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Medtronic Bifurcation Stent System
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 45
Region of Enrollment [Number; unit: participants]
  Australia | 39
  New Zealand | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Target Vessel Failure (TVF) at 30 Days Post Procedure.
Description: TVF was reported if any of the following events occurred: Recurrent MI in territory not clearly attributed to a vessel other than the target lesion; Cardiac death not clearly due to a non-target vessel endpoint or Clinically driven target revascularization.
Time Frame: 30 days
Measure: Number; unit: Participants
Arm/Group | Subjects Receiving Bifurcation Stents
Number analyzed (Participants) | 52
Participants | 2

2. Secondary Outcome: Device Success
Description: Device success is reported as Historical-standard definition: attainment of <50% residual stenosis of all target lesion/s using only the assigned device and any adjunct stents as specified in the Investigational Plan.
Time Frame: During index procedure
Population: ITT included all subjects after a run-in subject at each site.
Measure: Number; unit: participants
Arm/Group | Bifurcation Stent System
Number analyzed (Participants) | 53
participants | 46

3. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) at 6 Months
Description: as for outcome 1
Time Frame: 6 month
Population: Includes all patients receiving bifurcation stent and having evaluable data.
Measure: Number; unit: participants
Arm/Group | Bifurcation Stent System
Number analyzed (Participants) | 47
participants | 4

4. Secondary Outcome: Number of Participants With Target Vessel Failure at 9 Months.
Description: as for outcome 1
Time Frame: 9 month
Population: Includes all subjects receiving bifurcation stents and having evaluable data
Measure: Number; unit: participants
Groups:
- Bifurcation Stent System: Evaluable patients within pre-specified follow up window
Arm/Group | Bifurcation Stent System
Number analyzed (Participants) | 47
participants | 6

5. Secondary Outcome: Number of Participant With Target Vessel Failure at 12 Months
Description: as for outcome 1
Time Frame: 12 month
Population: Includes all subjects receiving bifurcation stents and having evaluable data.
Measure: Number; unit: participants
Arm/Group | Subjects Receiving Bifurcation Stents
Number analyzed (Participants) | 47
participants | 6

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- 1. Branch Bifurcation Stent System: All subjects enrolled in the BRANCH study
Arm/Group | 1. Branch Bifurcation Stent System
Serious Adverse Events (participants affected / at risk) | 23/60
Other Adverse Events (participants affected / at risk) | 46/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Branch Bifurcation Stent System (N=60)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Angina Pectoris (Cardiac disorders) | 8 (9)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 4 (4)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Visual Disturbance (Eye disorders) | 1 (1)
Chest Pain (General disorders) | 5 (6)
Non-Cardiac Chest Pain (General disorders) | 2 (2)
Device Malfunction (Injury, poisoning and procedural complications) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope Vasovagal (Nervous system disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Coronary Revascularisation (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Branch Bifurcation Stent System (N=60)
Bradycardia (Cardiac disorders) | 5 (5)
Coronary Artery Dissection (Cardiac disorders) | 8 (9)
Nausea (Gastrointestinal disorders) | 4 (4)
Chest Pain (General disorders) | 8 (10)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Syncope Vasovagal (Nervous system disorders) | 4 (4)
Haematoma (Vascular disorders) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less